CLINICAL TRIAL: NCT00428584
Title: A Randomized, Multicenter, Two Arm, Open Label, Twelve Week Phase IIIb Study to Evaluate the Tolerability of Rebif (New Formulation) (IFN Beta-1a) and Betaseron (IFN Beta-1b) in IFN-naive Subjects With Relapsing Remitting Multiple Sclerosis (RRMS) Followed by a Single Arm, Eighty-two Week Minimum, Rebif (New Formulation) Only Safety Extension
Brief Title: RNF and Betaseron® Tolerability Study
Acronym: REFORMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Fernando Dangond, EMD Serono
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27133
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Results first posted 2010-03-04 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Relapsing Remitting Multiple Sclerosis (RRMS)
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1b

ARMS (2):
- 1 (Experimental): interferon beta-1a
  Interventions: Drug: New Formulation of rebif - human interferon beta-1a
- 2 (Active Comparator): interferon beta-1b
  Interventions: Drug: Interferon beta -1b

INTERVENTIONS:
Drug: New Formulation of rebif - human interferon beta-1a — New Formulation of rebif- 44 mcg, SC (sub-cutaneous) thrice weekly (tiw) injection.
  Arms: 1
Drug: Interferon beta -1b — Betaseron - 250 mcg, SC (sub-cutaneous) every other day injection.
  Arms: 2

SUMMARY:
To evaluate the tolerability of a new formulation of rebif and Betaseron in subjects with relapsing-remitting multiple sclerosis (RRMS) by comparing the mean change in injection site pain scores from pre-injection to 30 minutes post therapy administration.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with diagnosis of RRMS according to McDonald criteria or Poser
2. Subject is between 18 and 60 years old inclusive
3. Subject is willing to follow study procedures
4. Subject has given written informed consent
5. Female subjects must be neither pregnant nor breast-feeding and must lack childbearing potential, as defined by either:

   * Being post-menopausal or surgically sterile, or
   * Using a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, or condom with spermicide, for the duration of the study.

Exclusion Criteria:

1. Subject has Clinically Isolated Syndrome (CIS), Primary Progressive MS, or Secondary Progressive MS without superimposed relapses.
2. Subject has had any prior interferon beta therapy (either beta-1b or beta-1a) prior to study Day 1.
3. Subject received any other approved disease modifying therapy for MS (glatiramer acetate) or any cytokine or anti-cytokine therapy within the 3 months prior to Study Day 1.
4. Subject received immunomodulatory or immunosuppressive therapy (including but not limited to cyclophosphamide, cyclosporin, methotrexate, azathioprine, linomide, mitoxantrone, teriflunomide, natalizumab, laquinimod, Campath and cladribine) within the 12 months prior to Study Day 1.
5. Subject had prior use of Cladribine or has previously received total lymphoid irradiation.
6. Subject has known allergy to natural or recombinant interferon or any other component of formulation excipient(s) of Rebif® or Betaseron®: Mannitol, Poloxamer 188, Methionine, Benzyl alcohol or Albumin (human).
7. Use of any other injectable medications on a regular basis during the week prior to the screening period or during the screening or treatment periods. Receiving a single injection for treatment or prophylaxis of a condition unrelated to the subject's multiple sclerosis or the subject's Rebif® or Betaseron® therapy (e.g. receiving a influenza or pneumococcus vaccination) is acceptable.
8. History of any chronic pain syndrome.
9. Subject has any other disease apart from MS that could better explain the subjects signs and symptoms.
10. Subject has complete transverse myelitis or bilateral optic neuritis.
11. Subjects who used any investigational drug or experimental procedure within 12 weeks prior to visit 1.
12. Subject has inadequate liver function, defined by a total bilirubin, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) or alkaline phosphatase > 2.5 times the upper limit of the normal values.
13. Subject has inadequate bone marrow reserve, defined as a white blood cell count less than 0.5 x lower limit of normal.
14. Subject suffers from current autoimmune disease (other than RRMS).
15. Subject suffers from major medical or psychiatric illness that in the opinion of the investigator creates undue risk to the subject or could affect compliance with the study protocol
16. Subject is pregnant or attempting to conceive
17. Visual or physical impairment that precludes completion of diaries and questionnaires.
18. Subject received oral or systemic corticosteroids or ACTH within 30 days of visit 1.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2006-12; Primary Completion 2007-11 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Dangond, MD, Study Director — EMD Serono
Locations (1):
- EMD Serono Med Info, Rockland, Massachusetts, United States

REFERENCES:
- [Derived] Singer B, Bandari D, Cascione M, LaGanke C, Huddlestone J, Bennett R, Dangond F; REFORMS Study Group. Comparative injection-site pain and tolerability of subcutaneous serum-free formulation of interferonbeta-1a versus subcutaneous interferonbeta-1b: results of the randomized, multicenter, Phase IIIb REFORMS study. BMC Neurol. 2012 Dec 6;12:154. doi: 10.1186/1471-2377-12-154. PMID 23216674
- See also: Full FDA approved prescribing information can be found here — http://www.mslifelines.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 129 subjects were recruited from 27 Multiple Sclerosis (MS) Clinics in the US from December 2006 through August 2007.
Pre-assignment Details: Subjects had a pre-study evaluation period (screening) within 14 days of Study Day 1 which consisted of informed consent, medical/disease history, physical exam and laboratory assessments.
Groups:
- New Formulation of Rebif: The new formulation of rebif is not approved and under investigation in the US
Period: Comparative Phase
Arm/Group | New Formulation of Rebif | Betaseron
Started | 65 | 64
Completed | 56 (Comparator Phase - new formulation of rebif and Betaseron) | 63
Not Completed | 9 | 1
Period: Extension Phase
Arm/Group | New Formulation of Rebif | Betaseron
Started | 56 (Extension Phase - new formulation of rebif to new formulation of rebif) | 63
Completed | 35 | 34
Not Completed | 21 | 29

BASELINE CHARACTERISTICS:
Groups:
- New Formulation of Rebif: Human interferon beta 1a, (new formulation of rebif) 44 mcg, subcutaneous injection, three times a week
- Betaseron: Human interferon beta-1b, Betaseron 250 mcg, subcutaneous injection, every other day
- Total: Total of all reporting groups
Arm/Group | New Formulation of Rebif | Betaseron | Total
Number analyzed (Participants) | 65 | 64 | 129
Age Continuous [Mean (Standard Deviation); unit: years] | 40.26 (9.80) | 40.78 (9.56) | 40.52 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 44 | 90
  Male | 19 | 20 | 39
Region of Enrollment [Number; unit: participants]
  United States | 65 | 64 | 129

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) of Patient Reported Pain: Change in Mean VAS for the 21 Full-dose Injections at Pre-injection and 30 Minutes Post-injection Timepoints
Description: Subject reported perception of pain on the VAS where the slash drawn by the patient represents pain of increasing intensity from 0 (no pain) to 100 (worse possible pain), measured in millimeters. Mean VAS of 21 injections for each patient at pre-injection compared to mean VAS of 21 injections for each patient 30 minutes post-injection
Time Frame: From pre-injection to 30 minutes post injection of the VAS pain scores across the first 21 injections of full dose therapy of a new formulation of rebif and Betaseron
Population: One subject from the new formulation of rebif group discontinued due to pregnancy therefore, data for the Full Dose Calculation 30min Mean Change was not calculated
Measure: Mean (Full Range); unit: mm
Arm/Group | New Formulation of Rebif | Betaseron
Number analyzed (Participants) | 64 | 64
mm
  Mean Pre-Injection VAS Score | 0.43 (2.06) [0 to 16.29] | 0.40 (1.64) [0 to 12.42]
  Mean VAS at 30 minutes Post-Injection | 1.10 (4.24) [0 to 32.9] | 1.54 (5.19) [0 to 38.32]
  Mean Change to 30 Minutes Post-Injection | 0.67 (2.32) [-.43 to 16.62] | 1.14 (4.81) [-.33 to 38.05]
Statistical Analysis 1: Comparison: New Formulation of Rebif vs Betaseron; The primary efficacy endpoint was analyzed by using a two-way ANOVA model on ranked data including treatment group and site as fixed effect; Test type: Superiority or Other; p = 0.524, ANOVA — P value refers to mean change to 30 minute post injection

2. Secondary Outcome: Change in Mean VAS for the 21 Full-dose Injections at Pre-injection and Immediately After Injection Timepoints
Description: A visual analog scale (VAS) ranging from 0 to 100 mm on which subjects rate pain from no pain (0 mm) to worst possible pain (100 mm) was used. Mean VAS of 21 injections for each patient at pre-injection compared to mean VAS of 21 injections for each patient immediately after injection.
Time Frame: Pre-Injection to Immediately after Injection
Population: One subject from the new formulation of rebif group discontinued due to pregnancy
Measure: Mean (Full Range); unit: millimeters
Arm/Group | New Formulation of Rebif | Betaseron
Number analyzed (Participants) | 64 | 64
millimeters | 1.46 (2.93) [-.53 to 17.62] | 4.63 (10.02) [-.10 to 54.86]
Statistical Analysis 1: Comparison: New Formulation of Rebif vs Betaseron; Test type: Superiority or Other; p = 0.484, ANOVA

3. Secondary Outcome: Change in Mean VAS for the 21 Full-dose Injections at Pre-injection and 10 Minutes Post-injection Timepoints
Description: A visual analog scale (VAS) ranging from 0 to 100 mm on which subjects rate pain from no pain (0 mm) to worst possible pain (100 mm) was used. Mean VAS of 21 injections for each patient at pre-injection compared to mean VAS of 21 injections for each patient 10 minutes post injection.
Time Frame: Pre-injection to 10 minutes post-injection
Population: One subject from the new formulation of Rebif group discontinued due to pregnancy
Measure: Mean (Full Range); unit: Millimeters
Arm/Group | New Formulation of Rebif | Betaseron
Number analyzed (Participants) | 64 | 64
Millimeters | 0.70 (1.89) [-.33 to 10.19] | 1.89 (5.45) [-.56 to 36.74]
Statistical Analysis 1: Comparison: New Formulation of Rebif vs Betaseron; Test type: Superiority or Other; p = 0.838, ANOVA

4. Secondary Outcome: Number of Pain Free Patients at 30 Minutes Post-injection
Description: A visual analog scale (VAS) ranging from 0 to 100 mm on which subjects rate pain from no pain (0 mm) to worst possible pain (100 mm) was used.
  Pain-free was defined as a VAS score of 0 for all 21 full-dose injections for the Intent-to-Treat (ITT) population.
Time Frame: 30 minutes post injection
Population: One subject from the new formulation of rebif group discontinued due to pregnancy
Measure: Number; unit: Participants
Arm/Group | New Formulation of Rebif | Betaseron
Number analyzed (Participants) | 64 | 64
Participants | 31 | 28
Statistical Analysis 1: Comparison: New Formulation of Rebif vs Betaseron; Test type: Superiority or Other; p = 0.451, Cochran-Mantel-Haenszel — No pain is defined as a VAS = 0 for all 21 full dose injections

5. Secondary Outcome: Diameter of Injection Site Redness
Description: Blinded assessment of mean change in diameter of redness (in mm) at an injection site following an injection
Time Frame: 1-72 hours post injection over the first 12 weeks including the titration period
Population: One subject from the new formulation of rebif group discontinued due to pregnancy
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | New Formulation of Rebif | Betaseron
Number analyzed (Participants) | 64 | 64
mm | 8.28 (9.51) | 6.87 (7.67)
Statistical Analysis 1: Comparison: New Formulation of Rebif vs Betaseron; Test type: Superiority or Other; p = 0.338, ANOVA

6. Other Pre Specified Outcome: Secondary Outcome - Extension Phase: Change in Mean (mm) VAS for Pre-injection and Immediately After Injection Timepoints
Description: as for outcome 2
Time Frame: Pre-injection and immediately after injection
Population: 3 subjects discontinued and withdrew consent from the Betaseron to the new formulation of rebif group in the Extension Phase
Measure: Mean (Full Range); unit: millimeters
Groups:
- New Formulation of Rebif: Human interferon beta 1a, new formualation of rebif- 44 mcg, subcutaneous injection, three times a week
- Betaseron to New Formulation of Rebif: Human interferon beta-1b, Betaseron 250 mcg, subcutaneous injection, every other day
Arm/Group | New Formulation of Rebif | Betaseron to New Formulation of Rebif
Number analyzed (Participants) | 55 | 58
millimeters | 1.67 [-0.10 to 19.18] | 2.50 [-0.18 to 40.75]

7. Other Pre Specified Outcome: Secondary Outcome - Extension Phase: Change in Mean VAS at Pre-injection and 10 Minutes Post Injection
Time Frame: Pre-injection and 10 minutes post injection
Population: as for outcome 6
Measure: Mean (Full Range); unit: Millimeters
Groups:
- New Formulation of Rebif: Human interferon beta 1a, Rebif (New Formulation) 44 mcg, subcutaneous injection, three times a week
Arm/Group | New Formulation of Rebif | Betaseron to the New Formulation of Rebif
Number analyzed (Participants) | 55 | 58
Millimeters | 0.40 [-2.09 to 10.00] | 0.91 [-0.15 to 16.30]

8. Other Pre Specified Outcome: Secondary Outcome - Extension Phase: Number of Pain Free Patients at 30 Minutes Post Injection
Time Frame: Pain free patients at 30 minutes post injection
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | New Formulation of Rebif | Betaseron to the New Formulation of Rebif
Number analyzed (Participants) | 55 | 58
Participants | 30 | 36

9. Other Pre Specified Outcome: Secondary Outcome - Extension Phase: Diameter in Injection Site Redness
Time Frame: 1 to 72 hours post injection
Population: 3 subjects discontinued and withdrew consent from the Betaseron to Rebif New Formulation Group in the Extension Phase
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | New Formulation of Rebif | Betaseron to the New Formulation of Rebif
Number analyzed (Participants) | 55 | 58
Millimeters | 10.79 (13.89) | 7.46 (10.57)

10. Other Pre Specified Outcome: Primary Outcome - Extension Phase: Visual Analog Scale (VAS) of Patients Reported Pain; Change in Mean VAS at Pre-injection and 30 Minutes Post Injection
Time Frame: Pre-injection and 30 minutes post injection
Population: as for outcome 6
Measure: Mean (Full Range); unit: Millimeters
Arm/Group | New Formulation of Rebif | Betaseron to the New Formulation of Rebif
Number analyzed (Participants) | 55 | 58
Millimeters | 0.34 [-0.55 to 5.36] | 0.42 [-1.17 to 9.79]

ADVERSE EVENTS:
Arm/Group | New Formulation of Rebif | Betaseron
Serious Adverse Events (participants affected / at risk) | 4/65 | 5/64
Other Adverse Events (participants affected / at risk) | 62/65 | 57/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | New Formulation of Rebif (N=65) | Betaseron (N=64)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis / gallstones (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chronic Hepatits (Hepatobiliary disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | New Formulation of Rebif (N=65) | Betaseron (N=64)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 3 (4) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal PainUpper (Gastrointestinal disorders) | 4 (4) | 2 (2)
Anaphylactic Reaction (Immune system disorders) | 1 (1) | 0 (0)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Chronic Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (5)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0)
Dental Caries (Gastrointestinal disorders) | 1 (3) | 0 (0)
Dental Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 7 (9)
Drug Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 2 (4) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (9)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Eustachian Tube Obstruction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eye Pain (Eye disorders) | 1 (1) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 3 (3)
General Disorders and Administration site condition (General disorders) | 44 (236) | 45 (244)
Gingival Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Halo Vision (Eye disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (3) | 1 (1)
Infections and Infestations (Infections and infestations) | 38 (98) | 33 (76)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 14 (35) | 10 (23)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Investigations (Investigations) | 28 (58) | 15 (21)
Iritis (Eye disorders) | 0 (0) | 1 (1)
Iron Defficiency Anamia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Lip Dry (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 4 (4) | 5 (6)
Middle Ear Effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Mouth Ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 28 (61) | 27 (83)
Nausea (Gastrointestinal disorders) | 9 (22) | 5 (9)
Nervous system disorders (Nervous system disorders) | 29 (150) | 29 (211)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Phychiatric (Psychiatric disorders) | 16 (25) | 25 (36)
Platelet Disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Renal Disorder (Renal and urinary disorders) | 5 (5) | 4 (5)
Reproductive system and breast disorder (Reproductive system and breast disorders) | 4 (4) | 4 (5)
Respiratory, thoracic and mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 14 (26) | 13 (26)
Skin disorders (Skin and subcutaneous tissue disorders) | 11 (16) | 11 (15)
Stomach Discomfort (Gastrointestinal disorders) | 2 (3) | 1 (2)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 3 (4)
Tongue Ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth Disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vascular disorders (Vascular disorders) | 4 (4) | 3 (14)
Vertigo (Ear and labyrinth disorders) | 4 (4) | 3 (3)
Vision Blurred (Eye disorders) | 0 (0) | 2 (4)
Visual Disturbance (Eye disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither Institution nor any Principal Investigators shall publish or present any results from such Study to any third parties until: (i) EMD Serono publishes the results from all sites participating in such Study; (ii) Institution receives notification from EMD Serono that publication of the multi-site results is no longer planned; or (iii) twenty-four (24) months following the completion of the multi-site study at all sites, whichever occurs first.